CLINICAL TRIAL: NCT02879175
Title: Patients' Follow-up After Subarachnoid Haemorrhage Caused by Ruptured Intracranial
Brief Title: Patients' Follow-up After Subarachnoid Haemorrhage Caused by Ruptured Intracranial Aneurysms
Acronym: FUSAC
Status: Active, not recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: RBC_2016_9
Record Dates: First submitted 2016-08-22; First posted 2016-08-25 (Estimated); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Intracranial Aneurysms
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
After endovascular treatment of the intracranial aneurysm, recanalization may occur, with a risk of recurrent subarachnoid haemorrhage or long-term angiographic recurrences of aneurysms.

Few data exist on patients' long-term follow-up after subarachnoid haemorrhage caused by ruptured intracranial aneurysms.

ELIGIBILITY:
Inclusion Criteria:

- Patient treated with embolization for SAH due to aneurysmal rupture

Exclusion Criteria:

- Patient refusal to participate in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing endovascular treatment for a subarachnoid haemorrhage caused by ruptured intracranial aneurysms.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2016-09-08 (Actual); Primary Completion 2031-09 (Estimated); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
early neurological clinical recovery | 1 year after Subarachnoid Haemorrhage
  modified Rankin scale

CONTACTS AND LOCATIONS:
Overall Officials: Raphaël BLANC, Principal Investigator — Fondation ophtalmologique de Rothschild
Locations (1):
- Fondation Opthalmologique A de Rothschild, Paris, France, France